CLINICAL TRIAL: NCT06438640
Title: Implementation and Evaluation of a Strategy to Improve Pre-Anesthesia Care Discussions (My Anesthesia Choice-Hip Fracture)
Brief Title: Evaluating a Strategy to Improve Pre-Anesthesia Care Discussions (My Anesthesia Choice-Hip Fracture)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Wake Forest University Health Sciences (Other); University of Florida (Other); Dartmouth-Hitchcock Medical Center (Other); Henry Ford Health System (Other); The Cleveland Clinic (Other); Dartmouth College (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 855203
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Hip Fractures; Femoral Neck Fractures; Intertrochanteric Fractures; Subtrochanteric Fractures
Keywords: hip fracture; femoral neck; intertrochanteric; subtrochanteric; fracture; anesthesia; observational study; survey; shared decision making; My Anesthesia Choice; MAC-HF
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care will be delivered at each site during the pre-intervention phase. Patients treated in this arm will undergo pre-anesthesia care discussions as per existing clinical routine at each site.
- My Anesthesia Choice- HF (Active Comparator): During the intervention and sustainment phases, site clinicians will receive standardized in-personal or virtual training on shared decision making theory and approaches. The My Anesthesia Choice-HF tool will be made available for use during preoperative conversations. Clinicians will receive encouragement to use the tool on study-eligible patients based on their assessment of clinical appropriateness.
  Interventions: Behavioral: My Anesthesia Choice-HF Model

INTERVENTIONS:
Behavioral: My Anesthesia Choice-HF Model — Brief clinician training on shared decision making, paired with provision of a 1-page tabular format conversation aid listing answers to frequently asked questions regarding common anesthesia options for hip fracture surgery (spinal anesthesia; general anesthesia)
  Arms: My Anesthesia Choice- HF

SUMMARY:
The objective of this study is to assess the implementation process for and the effectiveness of a quality improvement (QI) strategy to increase shared decision-making around anesthesia options for hip fracture surgery at 6 US hospitals. The QI strategy is to be facilitated by a clinician-administered 1-page bedside conversation aid designed to improve the quality of physician-patient communication, paired with brief clinician training. The evaluation will occur via a stepped wedge, cluster randomized trial to be carried out over a period of 27 months.

DETAILED DESCRIPTION:
The objective of this study is to assess the implementation process for and the effectiveness of a quality improvement (QI) strategy to increase shared decision-making around anesthesia options for hip fracture surgery at 6 US hospitals. The QI strategy is to be facilitated by a clinician-administered 1-page bedside conversation aid designed to improve the quality of physician-patient communication, paired with brief clinician training. The evaluation will occur via a stepped wedge, cluster randomized trial to be carried out over a period of 27 months.

Activities at each site will be divided into three phases: Pre-Implementation; Active Implementation; and Sustainment. Data collection will occur across all study phases at each site, although specific data elements collected will vary across phases. To facilitate evaluation, sites will be randomly assigned to one of three possible timing sequences (A, B, C) for project implementation (2 sites/sequence). The duration of the active implementation phase will be the same for each sequence (12 months); however, the duration of pre-implementation and sustainment phases will vary across sequences.

During the pre-implementation phase, data collection on selected outcome variables will occur but no interventions will be delivered. During the implementation phase, site clinicians will undergo training in use of the My Anesthesia Choice-HF tool and the tool will be made available for use in clinical areas with eligible patients. Data collection on key outcomes will continue over this period, and clinicians will receive reminders to encourage tool use. During Sustainment, the tool will remain available for use and outcomes will continue to be measured to assess sustainment of the intervention over time.

ELIGIBILITY:
Inclusion:

Age 50 and older Planned surgery to treat a hip fracture

Exclusion:

Contraindication to spinal anesthesia: current anticoagulant therapy or coagulopathy Contraindication to spinal anesthesia: critical aortic stenosis Contraindication to spinal anesthesia: skin infection over the lumbar spine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3548 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Intervention reach (primary implementation outcome) | Day of surgery
  Reach of the intervention will be assessed as the rate of use of the conversation aid during the active implementation phase at each site among eligible patients during the pre-anesthesia evaluation. Data will be collected during the implementation phase at each site.
Shared Decision-Making Process scale score (SDMP; primary effectiveness outcome) | Postoperative day 0-3
  SDMP is a 4-item measure of shared decision making; this will be assessed on eligible patients during the pre-implementation and implementation phases of the study to allow for comparison of scores among eligible patients treated in the two periods

SECONDARY OUTCOMES:
CollaboRATE shared decision making scale score (secondary effectiveness outcome). | Postoperative day 0-3
  A 3-item measure of shared decision making; this will be assessed on eligible patients during the pre-implementation and implementation phases of the study to allow for comparison of scores among eligible patients treated in the two periods

OTHER OUTCOMES:
Decisional conflict | Postoperative day 0-3
  The fraction of patients reporting decisional conflict about anesthesia pre-implementation versus active implementation periods will be assessed via the 4-item SURE measure.
Knowledge regarding anesthesia options | Postoperative day 0-3
  Patient-reported knowledge about anesthesia options during the pre-implementation versus active implementation periods will be assessed by a 6-item brief knowledge evaluation
Willingness to recommend anesthesia type | Postoperative day 0-3
  Patient satisfaction with anesthesia care during the pre-implementation versus active implementation periods will be assessed by a single-item "willingness to recommend to friends and family" satisfaction measure.
Anesthesia type received | Day of surgery
  The fraction of patients receiving general versus spinal anesthesia will be compared during the pre-implementation versus active implementation periods.
Recovery of ambulation | Postoperative day 30 to 90
  The fraction of patients who are able to ambulate independently (i.e. without human assistance) at first clinic follow up between 30 and 90 days after surgery will be compared during the pre-implementation versus implementation periods.
Fidelity of intervention delivery | Day of surgery
  Fidelity of implementation to recommended best practices during active implementation and sustainment phases, assessed via the 9-item UPFRONT Fidelity Assessment. This item will be assessed on approximately 10% of patients treated in each phase
Sustainment of intervention | Day of surgery
  The percentage of eligible patients receiving the strategy during the sustainment phase
Perceived sustainability of the intervention | Study months 12-27
  Study clinicians' perceptions regarding sustainability of the intervention will be assessed during the implementation and sustainment phases via the 23-item NoMAD sustainability assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Neuman, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - University of Florida Gainesville, Gainesville, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic-Fairview, Cleveland, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Goldstein EC, Politi MC, Baraldi JH, Elwyn G, Campos H, Feng R, Mehta S, Whatley K, Schmitz V, Neuman MD. Refining, implementing, and evaluating an anesthesia choice conversation aid for older adults with hip fracture: protocol for a stepped wedge cluster randomized trial. Implement Sci Commun. 2024 Sep 12;5(1):97. doi: 10.1186/s43058-024-00635-3. PMID 39267183